CLINICAL TRIAL: NCT02209181
Title: A Randomized, Double-blind, Placebo- and Active-controlled Trial to Investigate the Single-dose Efficacy, Safety, and Pharmacokinetics of 250 and 1000 mg JNJ-10450232 in Postoperative Dental Pain
Brief Title: A Dental Pain Study to Test the Effectiveness of a New Pain Reliever Medicine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO-131230135611-CTPA
Record Dates: First submitted 2014-07-22; First posted 2014-08-05 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Pain
Keywords: dental pain; post-surgical dental pain
MeSH Terms: conditions — Pain; Toothache | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- JNJ-10450232 250 mg (Experimental)
  Interventions: Drug: JNJ-10450232 / Not yet marketed
- JNJ-10450232 1000 mg (Experimental)
  Interventions: Drug: JNJ-10450232 / Not yet marketed
- Placebo (Placebo Comparator)
  Interventions: Drug: JNJ-10450232 / Not yet marketed
- Acetaminophen 1000 mg (Active Comparator)
  Interventions: Drug: acetaminophen / Tylenol

INTERVENTIONS:
Drug: JNJ-10450232 / Not yet marketed — Subjects who meet the randomization criteria at baseline within 4.5 hours after dental surgery will be assigned to one of four treatment groups stratified by pharmacokinetic blood sampling schedule and by baseline pain intensity level.
  Arms: JNJ-10450232 250 mg
Drug: JNJ-10450232 / Not yet marketed — Subjects who meet the randomization criteria at baseline within 4.5 hours after dental surgery will be assigned to one of four treatment groups stratified by pharmacokinetic blood sampling schedule and by baseline pain intensity level.
  Arms: JNJ-10450232 1000 mg
Drug: JNJ-10450232 / Not yet marketed — Subjects who meet the randomization criteria at baseline within 4.5 hours after dental surgery will be assigned to one of four treatment groups stratified by pharmacokinetic blood sampling schedule and by baseline pain intensity level.
  Arms: Placebo
Drug: acetaminophen / Tylenol — Subjects who meet the randomization criteria at baseline within 4.5 hours after dental surgery will be assigned to one of four treatment groups stratified by pharmacokinetic blood sampling schedule and by baseline pain intensity level.
  Arms: Acetaminophen 1000 mg

SUMMARY:
To assess the safety and effectiveness one dose of a new pain reliever medicine (JNJ-10450232 at either the 250 or 1000 mg strength) compared with placebo (sugar pill) or acetaminophen 1000 mg after surgical removal of third molars. The primary endpoint will evaluate pain relief effectiveness up to 6 hours after administration of the study drug.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo- and active-controlled, parallel group study to evaluate the efficacy, safety and pharmacokinetic profile of JNJ-10450232, administered as a single dose in capsules (250 or 1000 mg), over a 24 hour period after molar extractions. Subjects will stay at the research center for ~24 hours after administration of study drug. Healthy male subjects, ages 18 to 45 years inclusive, will be screened by medical history, vital signs, an electrocardiogram (ECG), and clinical laboratory tests. Eligible subjects will return to the clinic on the day of surgery and complete baseline vital signs and clinical laboratory tests. They will undergo dental extraction of a minimum of three third-molars and, if qualified, will be randomly assigned to one of four study treatments for pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-45 years
* At least moderate dental pain assessed by a categorical scale pain intensity scale and a score of at least 5 on the 11-point (0-10) pain intensity numerical rating scale (PI-NRS) following surgical removal of three third-molars

Exclusion Criteria:

* Subjects who are not otherwise healthy
* Test positive for the urine drug screen
* Taking prohibited medications will not be allowed to participate in this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 269 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Muse, MD, Principal Investigator — Jean Brown Research; Cathy Gelotte, Ph.D., Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Gelotte CK, Vakil AM, Zimmerman BA, Zannikos P, Mishra R, Eichenbaum G, Kuffner EK, Flores CM. JNJ-10450232 (NTM-006), A novel non-opioid with structural similarities to acetaminophen, produces relatively long-lasting analgesia after a single dose in patients undergoing 3rd molar extraction. Regul Toxicol Pharmacol. 2025 Sep;161 Suppl 1:105480. doi: 10.1016/j.yrtph.2023.105480. Epub 2023 Aug 23. PMID 37625518

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Three placebo capsules taken orally
- Acetaminophen 1000 mg: Two encapsulated 500 mg tablets and one placebo capsule taken orally
- JNJ-10450232 250 mg: One JNJ-10450232 250 mg capsule and two placebo capsules taken orally
- JNJ-10450232 1000 mg: One JNJ-10450232 250 mg capsule, one JNJ-10450232 750 mg capsule, and one placebo capsule taken orally
Period: Overall Study
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Started | 67 | 67 | 69 | 66
Completed | 66 | 66 | 68 | 66
Not Completed | 1 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg | Total
Number analyzed (Participants) | 67 | 67 | 69 | 66 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.2 (2.69) | 19.0 (1.64) | 19.0 (2.13) | 19.3 (1.95) | 19.1 (2.13)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 67 | 67 | 69 | 66 | 269
Region of Enrollment [Number; unit: participants]
  USA | 67 | 67 | 69 | 66 | 269

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Efficacy From 0 to 6 Hours After the Dose Using the Time-weighted Sum of Pain Intensity Difference (SPID 0-6)
Description: Time-weighted sum of pain intensity difference by first multiplying each pain intensity difference (PID) score by the time from the previous time point, and adding them together for each scheduled time point within 0-6 hours. Time points included 15 minutes, 30 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours. The minimum SPID 0-6 was -30 and the maximum SPID 0-6 was 60, where higher is better. Pain intensity is the amount of pain experienced on a scale of 1-10 (where 1=no pain and 10=very severe pain).
Time Frame: 6 Hours
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 4.37 (1.783) | 20.75 (1.783) | 8.95 (1.757) | 20.56 (1.797)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 16.38, 95% CI 2-sided [11.42 to 21.35], Standard Error of Mean 2.522
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.068, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 4.58, 95% CI 2-sided [-0.35 to 9.51], Standard Error of Mean 2.503
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 16.20, 95% CI 2-sided [11.21 to 21.18], Standard Error of Mean 2.531
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -11.81, 95% CI 2-sided [-16.73 to -6.88], Standard Error of Mean 2.503
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.941, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-5.17 to 4.80], Standard Error of Mean 2.531

2. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 15 Minutes Post Dose
Description: Pain intensity is the amount of pain experienced on a scale of 1-10 (where 1=no pain and 10=very severe pain). The PID will be derived by subtracting the pain intensity from the baseline pain intensity.
Time Frame: Baseline to 15 minutes post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.13 (0.11) | 0.25 (0.11) | 0.06 (0.11) | 0.21 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.448, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.12, 95% CI 2-sided [-0.19 to 0.42], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.618, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.08, 95% CI 2-sided [-0.38 to 0.22], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.621, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.08, 95% CI 2-sided [-0.23 to 0.38], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.207, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-0.49 to 0.11], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.794, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.04, 95% CI 2-sided [-0.34 to 0.26], Standard Error of Mean 0.15

3. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 30 Minutes Post Dose
Description: as for outcome 2
Time Frame: Baseline to 30 minutes post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.25 (0.19) | 1.59 (0.19) | 0.46 (0.18) | 0.71 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.34, 95% CI 2-sided [0.82 to 1.86], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.420, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.21, 95% CI 2-sided [-0.30 to 0.72], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.083, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.46, 95% CI 2-sided [-0.06 to 0.97], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.13, 95% CI 2-sided [-1.64 to -0.62], Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.88, 95% CI 2-sided [-1.40 to -0.37], Standard Error of Mean 0.26

4. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 45 Minutes Post Dose
Description: as for outcome 2
Time Frame: Baseline to 45 minutes post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.28 (0.24) | 3.22 (0.24) | 0.91 (0.23) | 1.51 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.93, 95% CI 2-sided [2.28 to 3.59], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.058, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.63, 95% CI 2-sided [-0.02 to 1.29], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.23, 95% CI 2-sided [0.57 to 1.89], Standard Error of Mean 0.34
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.30, 95% CI 2-sided [-2.96 to -1.65], Standard Error of Mean 0.33
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.71, 95% CI 2-sided [-2.37 to -1.04], Standard Error of Mean 0.34

5. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 1 Hour Post Dose
Description: as for outcome 2
Time Frame: Baseline to 1 hour post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.25 (0.26) | 3.98 (0.26) | 1.03 (0.26) | 2.19 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.73, 95% CI 2-sided [3.01 to 4.46], Standard Error of Mean 0.37
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.035, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.78, 95% CI 2-sided [0.06 to 1.49], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.94, 95% CI 2-sided [1.21 to 2.67], Standard Error of Mean 0.37
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.96, 95% CI 2-sided [-3.68 to -2.24], Standard Error of Mean 0.36
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.79, 95% CI 2-sided [-2.52 to -1.07], Standard Error of Mean 0.37

6. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 1.5 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 1.5 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.37 (0.28) | 4.35 (0.28) | 1.23 (0.28) | 2.85 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.99, 95% CI 2-sided [3.21 to 4.77], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.028, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.86, 95% CI 2-sided [0.09 to 1.64], Standard Error of Mean 0.39
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.48, 95% CI 2-sided [1.70 to 3.26], Standard Error of Mean 0.40
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -3.12, 95% CI 2-sided [-3.90 to -2.35], Standard Error of Mean 0.39
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.51, 95% CI 2-sided [-2.29 to -0.73], Standard Error of Mean 0.40

7. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 2 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 2 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.41 (0.31) | 4.20 (0.31) | 1.43 (0.31) | 3.48 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.78, 95% CI 2-sided [2.92 to 4.65], Standard Error of Mean 0.44
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.021, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.02, 95% CI 2-sided [0.16 to 1.88], Standard Error of Mean 0.44
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.06, 95% CI 2-sided [2.19 to 3.93], Standard Error of Mean 0.44
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.77, 95% CI 2-sided [-3.63 to -1.91], Standard Error of Mean 0.44
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.104, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.72, 95% CI 2-sided [-1.59 to 0.15], Standard Error of Mean 0.44

8. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 3 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 3 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.71 (0.34) | 3.84 (0.34) | 1.69 (0.34) | 3.86 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.13, 95% CI 2-sided [2.18 to 4.07], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.041, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.98, 95% CI 2-sided [0.04 to 1.92], Standard Error of Mean 0.48
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.14, 95% CI 2-sided [2.19 to 4.09], Standard Error of Mean 0.48
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.15, 95% CI 2-sided [-3.09 to -1.21], Standard Error of Mean 0.48
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.973, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.02, 95% CI 2-sided [-0.93 to 0.97], Standard Error of Mean 0.48

9. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 4 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 4 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.91 (0.36) | 3.78 (0.36) | 1.79 (0.35) | 4.17 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.87, 95% CI 2-sided [1.87 to 3.87], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.079, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.89, 95% CI 2-sided [-0.10 to 1.88], Standard Error of Mean 0.50
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.27, 95% CI 2-sided [2.27 to 4.27], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.99, 95% CI 2-sided [-2.98 to -1.00], Standard Error of Mean 0.50
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.440, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.39, 95% CI 2-sided [-0.61 to 1.40], Standard Error of Mean 0.51

10. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 5 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 5 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.01 (0.37) | 3.56 (0.37) | 1.82 (0.36) | 4.14 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.55, 95% CI 2-sided [1.52 to 3.57], Standard Error of Mean 0.52
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.118, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.81, 95% CI 2-sided [-0.21 to 1.83], Standard Error of Mean 0.52
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.13, 95% CI 2-sided [2.10 to 4.16], Standard Error of Mean 0.52
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.73, 95% CI 2-sided [-2.75 to -0.71], Standard Error of Mean 0.52
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.262, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.59, 95% CI 2-sided [-0.44 to 1.62], Standard Error of Mean 0.52

11. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 6 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 6 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.12 (0.37) | 3.04 (0.37) | 1.69 (0.37) | 4.07 (0.38)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.92, 95% CI 2-sided [0.88 to 2.96], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.271, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.58, 95% CI 2-sided [-0.45 to 1.61], Standard Error of Mean 0.52
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.95, 95% CI 2-sided [1.91 to 3.99], Standard Error of Mean 0.53
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.011, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.34, 95% CI 2-sided [-2.37 to -0.32], Standard Error of Mean 0.52
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.052, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.03, 95% CI 2-sided [-0.01 to 2.07], Standard Error of Mean 0.53

12. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 7 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 7 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.13 (0.37) | 2.38 (0.37) | 1.66 (0.37) | 3.94 (0.38)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.018, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.25, 95% CI 2-sided [0.21 to 2.29], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.310, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.53, 95% CI 2-sided [-0.50 to 1.56], Standard Error of Mean 0.52
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.80, 95% CI 2-sided [1.76 to 3.85], Standard Error of Mean 0.53
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.172, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.72, 95% CI 2-sided [-1.75 to 0.31], Standard Error of Mean 0.52
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.004, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.55, 95% CI 2-sided [0.51 to 2.60], Standard Error of Mean 0.53

13. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 8 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 8 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.15 (0.36) | 1.99 (0.36) | 1.51 (0.35) | 4.00 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.102, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.84, 95% CI 2-sided [-0.17 to 1.84], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.479, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.36, 95% CI 2-sided [-0.64 to 1.35], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.85, 95% CI 2-sided [1.85 to 3.86], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.345, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.48, 95% CI 2-sided [-1.47 to 0.52], Standard Error of Mean 0.51
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.01, 95% CI 2-sided [1.01 to 3.02], Standard Error of Mean 0.51

14. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 9 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 9 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.19 (0.36) | 1.69 (0.36) | 1.73 (0.36) | 3.91 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.338, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.49, 95% CI 2-sided [-0.52 to 1.51], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.299, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.53, 95% CI 2-sided [-0.47 to 1.54], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.72, 95% CI 2-sided [1.70 to 3.73], Standard Error of Mean 0.52
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.942, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.04, 95% CI 2-sided [-0.97 to 1.04], Standard Error of Mean 0.51
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.22, 95% CI 2-sided [1.21 to 3.24], Standard Error of Mean 0.52

15. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 10 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 10 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.08 (0.36) | 1.60 (0.36) | 1.57 (0.36) | 3.87 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.306, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.52, 95% CI 2-sided [-0.48 to 1.53], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.335, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.49, 95% CI 2-sided [-0.51 to 1.49], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.79, 95% CI 2-sided [1.78 to 3.80], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.946, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.03, 95% CI 2-sided [-1.03 to 0.97], Standard Error of Mean 0.51
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.27, 95% CI 2-sided [1.25 to 3.28], Standard Error of Mean 0.51

16. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 11 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 11 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.03 (0.36) | 1.58 (0.36) | 1.57 (0.36) | 3.70 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.279, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.55, 95% CI 2-sided [-0.45 to 1.56], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.292, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.54, 95% CI 2-sided [-0.46 to 1.53], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.67, 95% CI 2-sided [1.66 to 3.68], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.971, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.02, 95% CI 2-sided [-1.02 to 0.98], Standard Error of Mean 0.51
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.11, 95% CI 2-sided [1.11 to 3.12], Standard Error of Mean 0.51

17. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 12 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 12 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.08 (0.36) | 1.57 (0.36) | 1.39 (0.35) | 3.61 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.329, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.50, 95% CI 2-sided [-0.50 to 1.50], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.531, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.32, 95% CI 2-sided [-0.68 to 1.31], Standard Error of Mean 0.50
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.53, 95% CI 2-sided [1.53 to 3.54], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.722, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.18, 95% CI 2-sided [-1.17 to 0.81], Standard Error of Mean 0.50
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.04, 95% CI 2-sided [1.03 to 3.04], Standard Error of Mean 0.51

18. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 16 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 16 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.93 (0.35) | 1.37 (0.35) | 1.08 (0.35) | 3.43 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.380, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.44, 95% CI 2-sided [-0.54 to 1.42], Standard Error of Mean 0.50
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.767, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.15, 95% CI 2-sided [-0.83 to 1.12], Standard Error of Mean 0.49
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.50, 95% CI 2-sided [1.52 to 3.49], Standard Error of Mean 0.50
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.557, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.29, 95% CI 2-sided [-1.27 to 0.68], Standard Error of Mean 0.49
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.06, 95% CI 2-sided [1.08 to 3.05], Standard Error of Mean 0.50

19. Secondary Outcome: Pain Intensity Difference From Baseline (PID) Scores at 24 Hours Post Dose
Description: as for outcome 2
Time Frame: Baseline to 24 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.15 (0.39) | 1.41 (0.39) | 1.29 (0.38) | 3.47 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.640, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.26, 95% CI 2-sided [-0.83 to 1.35], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.798, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.14, 95% CI 2-sided [-0.94 to 1.22], Standard Error of Mean 0.55
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.32, 95% CI 2-sided [1.23 to 3.42], Standard Error of Mean 0.55
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.829, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.12, 95% CI 2-sided [-1.20 to 0.96], Standard Error of Mean 0.55
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.06, 95% CI 2-sided [0.97 to 3.16], Standard Error of Mean 0.55

20. Secondary Outcome: Pain Relief (PAR) Scores at 15 Minutes Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 15 minutes post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.27 (0.11) | 0.52 (0.11) | 0.33 (0.11) | 0.38 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.117, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.25, 95% CI 2-sided [-0.06 to 0.57], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.687, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.06, 95% CI 2-sided [-0.25 to 0.38], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.497, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.11, 95% CI 2-sided [-0.21 to 0.43], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.239, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-0.51 to 0.13], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.376, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.14, 95% CI 2-sided [-0.46 to 0.18], Standard Error of Mean 0.16

21. Secondary Outcome: Pain Relief (PAR) Scores at 30 Minutes Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 30 minutes post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.60 (0.23) | 2.38 (0.23) | 0.90 (0.23) | 1.03 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.78, 95% CI 2-sided [1.14 to 2.42], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.350, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.30, 95% CI 2-sided [-0.33 to 0.94], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.183, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.43, 95% CI 2-sided [-0.21 to 1.08], Standard Error of Mean 0.33
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.48, 95% CI 2-sided [-2.11 to -0.84], Standard Error of Mean 0.32
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.34, 95% CI 2-sided [-1.98 to -0.70], Standard Error of Mean 0.33

22. Secondary Outcome: Pain Relief (PAR) Scores at 45 Minutes Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 45 minutes post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.64 (0.30) | 4.42 (0.30) | 1.52 (0.30) | 2.11 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.78, 95% CI 2-sided [2.94 to 4.61], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.037, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.88, 95% CI 2-sided [0.05 to 1.71], Standard Error of Mean 0.42
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.47, 95% CI 2-sided [0.63 to 2.30], Standard Error of Mean 0.43
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.90, 95% CI 2-sided [-3.73 to -2.07], Standard Error of Mean 0.42
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.31, 95% CI 2-sided [-3.15 to -1.47], Standard Error of Mean 0.43

23. Secondary Outcome: Pain Relief (PAR) Scores at 1 Hour Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 1 hour post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 0.84 (0.33) | 5.18 (0.33) | 1.68 (0.32) | 3.09 (0.33)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 4.34, 95% CI 2-sided [3.43 to 5.25], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.067, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.85, 95% CI 2-sided [-0.06 to 1.75], Standard Error of Mean 0.46
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.26, 95% CI 2-sided [1.34 to 3.17], Standard Error of Mean 0.46
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -3.49, 95% CI 2-sided [-4.40 to -2.59], Standard Error of Mean 0.46
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.08, 95% CI 2-sided [-3.00 to -1.17], Standard Error of Mean 0.46

24. Secondary Outcome: Pain Relief (PAR) Scores at 1.5 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 1.5 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.01 (0.35) | 5.88 (0.35) | 2.13 (0.34) | 3.97 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 4.87, 95% CI 2-sided [3.90 to 5.84], Standard Error of Mean 0.49
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.023, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.13, 95% CI 2-sided [0.16 to 2.09], Standard Error of Mean 0.49
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.96, 95% CI 2-sided [1.98 to 3.93], Standard Error of Mean 0.50
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -3.75, 95% CI 2-sided [-4.71 to -2.78], Standard Error of Mean 0.49
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.91, 95% CI 2-sided [-2.89 to -0.94], Standard Error of Mean 0.50

25. Secondary Outcome: Pain Relief (PAR) Scores at 2 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 2 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.17 (0.38) | 5.88 (0.38) | 2.53 (0.38) | 4.90 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 4.71, 95% CI 2-sided [3.64 to 5.78], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.012, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.36, 95% CI 2-sided [0.30 to 2.42], Standard Error of Mean 0.54
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.73, 95% CI 2-sided [2.66 to 4.81], Standard Error of Mean 0.54
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -3.35, 95% CI 2-sided [-4.41 to -2.29], Standard Error of Mean 0.54
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.074, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.98, 95% CI 2-sided [-2.05 to 0.09], Standard Error of Mean 0.54

26. Secondary Outcome: Pain Relief (PAR) Scores at 3 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 3 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.59 (0.42) | 5.39 (0.42) | 2.90 (0.41) | 5.40 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.80, 95% CI 2-sided [2.63 to 4.97], Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.026, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.32, 95% CI 2-sided [0.16 to 2.48], Standard Error of Mean 0.59
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.82, 95% CI 2-sided [2.64 to 4.99], Standard Error of Mean 0.60
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.48, 95% CI 2-sided [-3.64 to -1.32], Standard Error of Mean 0.59
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.978, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.02, 95% CI 2-sided [-1.16 to 1.19], Standard Error of Mean 0.60

27. Secondary Outcome: Pain Relief (PAR) Scores at 4 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 4 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 1.92 (0.44) | 5.31 (0.44) | 2.99 (0.43) | 5.83 (0.44)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.40, 95% CI 2-sided [2.18 to 4.62], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.081, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.07, 95% CI 2-sided [-0.13 to 2.28], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.91, 95% CI 2-sided [2.69 to 5.14], Standard Error of Mean 0.62
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -2.32, 95% CI 2-sided [-3.53 to -1.11], Standard Error of Mean 0.61
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.407, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.52, 95% CI 2-sided [-0.71 to 1.74], Standard Error of Mean 0.62

28. Secondary Outcome: Pain Relief (PAR) Scores at 5 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 5 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.17 (0.45) | 5.00 (0.45) | 3.05 (0.45) | 5.77 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.83, 95% CI 2-sided [1.56 to 4.10], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.170, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.88, 95% CI 2-sided [-0.38 to 2.14], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.60, 95% CI 2-sided [2.33 to 4.87], Standard Error of Mean 0.65
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.95, 95% CI 2-sided [-3.21 to -0.69], Standard Error of Mean 0.64
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.235, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.77, 95% CI 2-sided [-0.50 to 2.04], Standard Error of Mean 0.65

29. Secondary Outcome: Pain Relief (PAR) Scores at 6 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 6 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.32 (0.46) | 4.42 (0.46) | 2.92 (0.45) | 5.68 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.10, 95% CI 2-sided [0.82 to 3.39], Standard Error of Mean 0.65
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.355, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.60, 95% CI 2-sided [-0.68 to 1.87], Standard Error of Mean 0.65
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.36, 95% CI 2-sided [2.07 to 4.65], Standard Error of Mean 0.65
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.021, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.50, 95% CI 2-sided [-2.78 to -0.23], Standard Error of Mean 0.65
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.056, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.26, 95% CI 2-sided [-0.03 to 2.55], Standard Error of Mean 0.65

30. Secondary Outcome: Pain Relief (PAR) Scores at 7 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 7 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.41 (0.46) | 3.62 (0.47) | 2.80 (0.46) | 5.57 (0.47)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.067, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.21, 95% CI 2-sided [-0.09 to 2.50], Standard Error of Mean 0.66
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.547, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.39, 95% CI 2-sided [-0.89 to 1.68], Standard Error of Mean 0.65
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.16, 95% CI 2-sided [1.86 to 4.46], Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.214, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.81, 95% CI 2-sided [-2.10 to 0.47], Standard Error of Mean 0.65
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.003, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.96, 95% CI 2-sided [0.66 to 3.26], Standard Error of Mean 0.66

31. Secondary Outcome: Pain Relief (PAR) Scores at 8 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 8 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.41 (0.45) | 3.10 (0.45) | 2.63 (0.44) | 5.62 (0.45)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.281, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.69, 95% CI 2-sided [-0.57 to 1.95], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.729, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.22, 95% CI 2-sided [-1.03 to 1.47], Standard Error of Mean 0.63
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.21, 95% CI 2-sided [1.95 to 4.47], Standard Error of Mean 0.64
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.459, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.47, 95% CI 2-sided [-1.72 to 0.78], Standard Error of Mean 0.63
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.52, 95% CI 2-sided [1.26 to 3.78], Standard Error of Mean 0.64

32. Secondary Outcome: Pain Relief (PAR) Scores at 9 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 9 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.46 (0.46) | 2.73 (0.46) | 2.98 (0.45) | 5.50 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.674, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.27, 95% CI 2-sided [-1.00 to 1.55], Standard Error of Mean 0.65
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.417, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.52, 95% CI 2-sided [-0.74 to 1.79], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.05, 95% CI 2-sided [1.77 to 4.33], Standard Error of Mean 0.65
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.698, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.25, 95% CI 2-sided [-1.02 to 1.52], Standard Error of Mean 0.64
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.77, 95% CI 2-sided [1.49 to 4.05], Standard Error of Mean 0.65

33. Secondary Outcome: Pain Relief (PAR) Scores at 10 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 10 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.28 (0.46) | 2.67 (0.46) | 2.81 (0.45) | 5.40 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.541, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.39, 95% CI 2-sided [-0.87 to 1.66], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.409, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.53, 95% CI 2-sided [-0.73 to 1.79], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 3.12, 95% CI 2-sided [1.85 to 4.39], Standard Error of Mean 0.65
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.834, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.13, 95% CI 2-sided [-1.12 to 1.39], Standard Error of Mean 0.64
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.73, 95% CI 2-sided [1.45 to 4.00], Standard Error of Mean 0.65

34. Secondary Outcome: Pain Relief (PAR) Scores at 11 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 11 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.26 (0.45) | 2.63 (0.45) | 2.75 (0.45) | 5.25 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.573, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.36, 95% CI 2-sided [-0.90 to 1.63], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.448, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.49, 95% CI 2-sided [-0.77 to 1.74], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.98, 95% CI 2-sided [1.71 to 4.25], Standard Error of Mean 0.64
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.848, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.12, 95% CI 2-sided [-1.13 to 1.38], Standard Error of Mean 0.64
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.62, 95% CI 2-sided [1.35 to 3.89], Standard Error of Mean 0.64

35. Secondary Outcome: Pain Relief (PAR) Scores at 12 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 12 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.34 (0.46) | 2.57 (0.46) | 2.53 (0.45) | 5.16 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.720, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.23, 95% CI 2-sided [-1.04 to 1.50], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.763, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.19, 95% CI 2-sided [-1.07 to 1.45], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.82, 95% CI 2-sided [1.55 to 4.09], Standard Error of Mean 0.65
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.952, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.04, 95% CI 2-sided [-1.30 to 1.22], Standard Error of Mean 0.64
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.59, 95% CI 2-sided [1.31 to 3.86], Standard Error of Mean 0.65

36. Secondary Outcome: Pain Relief (PAR) Scores at 16 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 16 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.09 (0.45) | 2.23 (0.45) | 2.07 (0.44) | 4.96 (0.45)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.821, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.14, 95% CI 2-sided [-1.10 to 1.39], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.978, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.02, 95% CI 2-sided [-1.25 to 1.22], Standard Error of Mean 0.63
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.88, 95% CI 2-sided [1.63 to 4.13], Standard Error of Mean 0.63
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.799, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.16, 95% CI 2-sided [-1.39 to 1.07], Standard Error of Mean 0.63
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.73, 95% CI 2-sided [1.49 to 3.98], Standard Error of Mean 0.63

37. Secondary Outcome: Pain Relief (PAR) Scores at 24 Hours Post Dose
Description: Pain relief is the amount of pain relief on a scale of 1-10 (where 1=no relief and 10=complete relief).
Time Frame: 24 hours post dose
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
units on a scale | 2.44 (0.49) | 2.20 (0.50) | 2.33 (0.49) | 4.96 (0.50)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.726, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.25, 95% CI 2-sided [-1.62 to 1.13], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.869, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.11, 95% CI 2-sided [-1.48 to 1.25], Standard Error of Mean 0.69
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.52, 95% CI 2-sided [1.13 to 3.90], Standard Error of Mean 0.70
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.851, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.13, 95% CI 2-sided [-1.24 to 1.50], Standard Error of Mean 0.69
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 2.76, 95% CI 2-sided [1.38 to 4.15], Standard Error of Mean 0.70

38. Secondary Outcome: Duration of Pain Relief After Dosing (Time to Rescue Medication)
Description: Time (minutes) to rescue medication was measured as the elapsed time from when the investigational product was given until the time rescue medication was given.
Time Frame: Completed at time of the first rescue medication (hours post dose), estimated up through Day 2
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
minutes | 109.0 [97.0 to 189.0] | 468.5 [370.0 to 607.0] | 129.0 [100.0 to 725.0] | NA [768.0 to NA] — Median and upper limit of the confidence interval were not estimable since less than 50% of the subjects treated with JNJ-10450232 1000 mg used rescue medication.
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups. Subjects who withdrew from the study before 24 hours, but did not use rescue therapy, were censored at the time of discontinuation. Subjects who did not rescue medication during the 24-hour study period had their time to rescue set to 24 hours and were censored at 24 hours; Test type: Superiority or Other; p = 0.042, Log Rank — The significance threshold level was 0.05 (two-sided). P-Value is from Log-rank test comparing survival curves
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; [analysis description as in outcome 38, analysis 1]; Test type: Superiority or Other; p = 0.779, Log Rank — The significance threshold level was 0.05 (two-sided). P-Value is from Log-rank test comparing survival curves
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; [analysis description as in outcome 38, analysis 1]; Test type: Superiority or Other; p < 0.001, Log Rank — The significance threshold level was 0.05 (two-sided). P-Value is from Log-rank test comparing survival curves
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; [analysis description as in outcome 38, analysis 1]; Test type: Superiority or Other; p = 0.196, Log Rank — The significance threshold level was 0.05 (two-sided). P-Value is from Log-rank test comparing survival curves
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; [analysis description as in outcome 38, analysis 1]; Test type: Superiority or Other; p = 0.006, Log Rank — The significance threshold level was 0.05 (two-sided). P-Value is from Log-rank test comparing survival curves

39. Secondary Outcome: Subject Global Evaluation
Description: How the subject would rate the study medication as a pain-reliever on a scale of 0-4 (where 0=poor and 4=excellent).
Time Frame: Completed at hour 12 or at time of the first rescue medication (hours post dose).
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Number analyzed (Participants) | 67 | 67 | 69 | 66
percentage of participants
  Poor (0) | 62.7 | 12.1 | 55.1 | 28.8
  Fair (1) | 14.9 | 9.1 | 4.3 | 6.1
  Good (2) | 11.9 | 30.3 | 21.7 | 22.7
  Very Good (3) | 10.4 | 42.4 | 15.9 | 30.3
  Excellent (4) | 0.0 | 6.1 | 2.9 | 12.1
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.5, 95% CI 2-sided [1.1 to 1.9], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.077, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 0.4, 95% CI 2-sided [-0.0 to 0.8], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 1.2, 95% CI 2-sided [0.8 to 1.6], Standard Error of Mean 0.21
Statistical Analysis 4: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 250 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-1.6 to -0.7], Standard Error of Mean 0.21
Statistical Analysis 5: Comparison: Acetaminophen 1000 mg vs JNJ-10450232 1000 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.148, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.21

ADVERSE EVENTS:
Time Frame: Within 7 days after dental surgery, +30 days for serious adverse events.
Description: Adverse events (AEs) were systematically collected during the study and during the adverse event follow-up telephone interview within 7 days after dental surgery. Serious AEs were reported through 30 days after product use. Spontaneously reported AEs collected outside of the regularly scheduled telephone interviews were also recorded. Any clinically important abnormalities or causally-related AEs events persisting were followed until resolution or until reaching a clinically stable endpoint.
Arm/Group | Placebo | Acetaminophen 1000 mg | JNJ-10450232 250 mg | JNJ-10450232 1000 mg
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/69 | 0/66
Other Adverse Events (participants affected / at risk) | 3/67 | 5/67 | 3/69 | 5/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | Acetaminophen 1000 mg (N=67) | JNJ-10450232 250 mg (N=69) | JNJ-10450232 1000 mg (N=66)
Blood Bilirubin Increased (Investigations) | 3 | 5 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less